CLINICAL TRIAL: NCT07231120
Title: A Phase I Clinical Study Evaluating the Safety, Tolerability, Pharmacokinetic Characteristics, and Preliminary Efficacy of SXRN Injection in Patients With Cancer Cachexia
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu Nutai Biologics Co., Ltd (Industry)
Collaborators: Jiangsu GQ Pharma Co., Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AA0102
Record Dates: First submitted 2025-09-23; First posted 2025-11-17 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-11

CONDITIONS: Cachexia-Anorexia Syndrome; Solid Tumor Malignancies
Keywords: cancer patient with anorexia-cachexia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SXRN (Experimental): Phase Ia: 3~4 dose cohorts are initially formulated, namely: 4 mg, 6mg, 8mg, and Xmg of SXRN Injection, utilizing the conventional "3+3" design for dose escalation. Participants will be enrolled sequentially into the 3~4 dose cohorts, starting from low to high.
  Phase Ib: 2 dose cohorts of SXRN Injection (tentatively 6 mg and 8 mg, based on phase Ia data) are initially formulated, in patients with cancers including but not limited to pancreatic cancer, non-small cell lung cancer, and colon cancer. Treatment will combine the standard anti-tumor therapy with SXRN Injection.
  The infusion on the first day for each dose cohort is referred to as C1D1, with the administration qd for 5 consecutive days, followed by a 2-day break; Each treatment cycle spans 3 weeks (21 days).
  The study plans to enroll 12-24 participants for phase Ia and 20-30 participants for phase Ib, and will be conducted at 1-2 center(s) nationwide.
  Interventions: Drug: SXRN Injection

INTERVENTIONS:
Drug: SXRN Injection — Intravenous infusion, qd for 5 consecutive days, followed by a 2-day break; every 3 weeks (21days) makes a treatment cycle. Ⅰa phase：conventional "3+3" design for dose escalation； Ⅰb phase：standard anti-tumor therapy combined with SXRN Injection

SUMMARY:
This is a clinical study evaluating the safety, tolerability, pharmacokinetics (PK), and preliminary efficacy of SXRN Injection in cancer patients with anorexia-cachexia. Phase Ia employs a single-arm, open-label, dose-escalation design. Phase Ib, an extension of the study, utilizes a design of combination therapy with standard anti-tumor therapy for cancers including but not limited to pancreatic cancer, non-small cell lung cancer (NSCLC), and colon cancer.

DETAILED DESCRIPTION:
This study is collaboratively sponsored by Jiangsu Nutai Biologics Co., Ltd. and Jiangsu GQ Co., Ltd.. Nutai serves as the Responsible Party for this registration.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all the following criteria for inclusion:

* 1. Male or female, aged 18 to 75 years (inclusive) at the time of signing the informed consent form (ICF);
* 2. Patients with histologically or cytologically confirmed advanced solid tumors, with at least one measurable or evaluable lesion according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1;
* 3. Diagnosed of cancer anorexia-cachexia based on the 2025 Guidelines for the Diagnosis and Treatment of Cancer Anorexia-Cachexia Syndrome and referring to Chinese population characteristics, i.e., meeting the following criteria (either ① + ② or ① + ③):

  ① >5% involuntary weight loss within the past 6 months; or >2% weight loss if BMI <18.5 kg/m²; or >2% weight loss in the presence of reduced muscle mass;

  ② Anorexia (VAS score ≤70, or FAACT-A/CS score ≤37);

  ③ CRP >5 mg/L;
* 4. (Phase Ia only) Cancer patients who have failed or are intolerant (experienced drug-related ≥ Grade 4 hematologic toxicity, or ≥ Grade 3 non-hematologic toxicity) to prior standard therapy, or lack effective conventional treatment options;
* 5. (Phase Ib only) Patients requiring standard anti-tumor drug therapy per CSCO guidelines of advanced pancreatic cancer, non-small cell lung cancer, colorectal cancer, or other eligible solid tumors;
* 6. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2;
* 7. Life expectancy ≥12 weeks.
* 8. Laboratory test results and organ function assessed within 7 days prior to the first dose must meet the following criteria:
* Blood routine: 1)Absolute Neutrophil Count (ANC) ≥1.5×10^9/L;2)Platlets (PLT) Count≥75×10^9/L; 3)Hemoglobins (Hb) ≥80 g/L.

Note: the criteria above shall still be maintained within 14 days before the initial infusion, either without the need of blood transfusion, or using supportive treatment including granulocyte colony-stimulating factor (G-CSF), thrombopoietin (TPO), interleukin-11 (IL-11), and erythropoietin (EPO), and etc.

* Blood biochemistry: 1)Total bilirubin (TBIL) ≤3.0 × upper limit of normal (ULN); 2)Serum creatinine (SCr) ≤1.5 × ULN or creatinine clearance (CrCl) by Cockroft Gault formula ≥30 mL/min; 3)Aspartate Amino Transferase (AST), Alanine Aminotransferase (ALT) ≤3×ULN; for participants with liver metastasis, AST, ALT≤5.0×ULN, and ALP≤6.0×ULN; d)Albumin (ALB) ≥30g/L.
* Urine routines: Urine protein ≤2+ (if >2+, 24-hour urine protein quantification must be performed, and total protein ≤1 g is required for eligibility).
* Blood coagulation: International Normalized Ratio (INR), Prothrombin Time (PT), Activated Partial Thromboplastin Time (APTT) ≤1.5×ULN.

Note: for subjects receiving precautious anti-coagulation treatment, the investigator shall determine whether INR and APTT remains in a safe and effective range for treatment.

* Ultrasonic cardiogram: Left Ventricular Ejection Fraction (LVEF) ≥50%.
* 9.The participant must be able to understand and voluntarily sign the written Informed Consent Form (ICF); and must be willing and able to comply with all study procedures and follow-up examinations.

Exclusion Criteria:

Participants meeting any of the following criteria shall be excluded from the study:

* 1. Reversible causes of reduced food intake as determined by the investigator, which may include but are not limited to mechanical obstruction preventing adequate oral intake;
* 2. Use of any prescription medication intended to improve appetite or mitigate weight loss within 28 days or 5 half-lives of the drug (whichever is shorter) prior to the first dose of the investigational product, including but not limited to anamorelin, megestrol acetate, cannabinoids, or medical marijuana;
* 3. Patients currently receiving tube feeding or parenteral nutrition support;
* 4. Treatment with any other investigational drug within 4 weeks or 5 half-lives (whichever is shorter) prior to the first dose of the study drug;
* 5. Patients with cachexia clearly attributable to other underlying conditions, such as severe chronic obstructive pulmonary disease (COPD), AIDS, etc.;
* 6. Hormonal therapy judged by the investigator as potentially to improve the assessment of cachexia-related outcomes.
* 7. Patients who have undergone major surgery or interventional procedures within 4 weeks prior to the first dose, or who are scheduled to undergo such procedures during the trial (excluding tumor biopsy, puncture, etc.);
* 8. Patients with toxicities from previous antitumor therapies that have not yet recovered to ≤ Grade 1 or baseline levels (except for toxicities judged by the investigator as to pose no safety risk, such as alopecia, or asymptomatic hypothyroidism induced by immune checkpoint inhibitors that is stable and only requires thyroid hormone replacement therapy);
* 9. Clinically uncontrolled third-space fluid accumulation (e.g., pleural effusion, ascites, or pericardial effusion), meeting any of the following criteria: moderate or larger volume, received local treatment (including drainage, peritoneal shunt, or cell-free concentrated ascites reinfusion therapy, etc.) within 2 weeks before screening or scheduled within the next 2 weeks, significant re-accumulation within 2 weeks after local treatment, or requiring long-term catheterization; or judged by the investigator as unsuitable for enrollment;
* 10.Patients with central nervous system metastases requiring intervention;
* 11.History of other malignancies, except for those who have undergone curative treatment with no recurrence within 5 years (e.g., carcinoma in situ of the cervix, basal cell carcinoma of the skin, etc.);
* 12.History of immunodeficiency, including acquired or congenital immunodeficiency diseases, organ transplantation, allogeneic bone marrow transplantation, or autologous hematopoietic stem cell transplantation;
* 13.(Non-infectious) pulmonary inflammation/interstitial lung disease requiring steroid therapy within 4 weeks prior to the first infusion;
* 14.History of severe cardiovascular or cerebrovascular diseases, including but not limited to:

  1. Severe cardiac rhythm or conduction abnormalities, such as ventricular arrhythmias requiring clinical intervention, second- or third-degree atrioventricular block, etc.;
  2. Cardiac dysfunction classified as Class III-IV per the New York Heart Association (NYHA) criteria;
  3. Acute coronary syndrome, congestive heart failure, aortic dissection, stroke, or other Grade 3 or higher cardiovascular/cerebrovascular events within 6 months prior to the first dose;
* 15.Hypertension uncontrolled by a stable regimen of antihypertensive medication (systolic blood pressure ≥160 mmHg, and/or diastolic blood pressure ≥100 mmHg);
* 16.Active chronic hepatitis B (e.g., HBsAg positive or HBcAb positive with HBV DNA above the lower limit of detection), active hepatitis C (e.g., HCV antibody positive with HCV RNA above the lower limit of detection), or human immunodeficiency virus (HIV) infection;
* 17.Active infection requiring systemic therapy within 2 weeks prior to the first dose;
* 18.History of active tuberculosis infection within 1 year prior to the first dose;
* 19.Any other uncontrolled or significant comorbid disease(s), either currently or historically, that by the investigator's judgment may interfere with trial participation or evaluation;
* 20.Known allergy or contraindication to the investigational product (SXRN injection) or its drug substance process-related impurities (e.g., spectinomycin);
* 21.For premenopausal female participants (postmenopausal females must be amenorrheic for at least 12 months to be considered of non-childbearing potential): serum pregnancy test as positive, or participants of childbearing potential (including female partners of male participants) who, in the investigator's opinion, are likely to become pregnant, are breastfeeding, or are unwilling to use effective contraception during the study and for at least 6 months after the last dose of the investigational product;
* 22. Any other condition that considered by the investigator as to render the patient unsuitable for participation in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2025-11-17 (Actual); Primary Completion 2026-11-09 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Phase Ia: MTD | Up to 90 days post last dosing
  To determine the Maximum Tolerated Dose (MTD) of SXRN Injection for the treatment of caner anorexia-cachexia.
Phase Ia&Ib: Incidence of Dose Limiting Toxicities (DLTs) | Up to 21 days after the first dosing of SXRN Injection for each patient
Phase Ib: RP2D | Up to 90 days post last dosing
  To determine the Recommended Phase II Dose (RP2D) of SXRN Injection.

SECONDARY OUTCOMES:
Maximum serum concentration (Cmax) of SXRN Injection; | Up to 90 days after the last dosing of SXRN Injection
Time to Cmax (Tmax) of SXRN Injection | Up to 90 days after the last dosing of SXRN Injection
Area under the curve from time "0" to the time of the last measurable concentration (AUC0-t) of SXRN Injection | Up to 90 days after the last dosing of SXRN Injection
Phase Ia&Ib: Average change in the severity of anorexia (based on the Functional Assessment of Anorexia/Cachexia Therapy - Anorexia/Cachexia Subscale-12 [FAACT-A/CS-12]) in the first cycle from baseline to each assessment timepoint. | Within 24 weeks from baseline
Phase Ia&Ib: Average change in quality of life (based on the EORTC Quality of Life Questionnaire [QLQ-C30]) in the first cycle from baseline to each assessment timepoint. | Within 24 weeks from baseline
Phase Ia&Ib: Average changes in comprehensive physical function (based on the 6-minute walk test [6MWT]) from baseline to each assessment timepoint. | Within 24 weeks from baseline
Phase Ia&Ib: Average change in body weight/lean body mass(LBM) from baseline to each assessment timepoint | Within 24 weeks from baseline
Overall sunvival (OS) | 12 months
progression free survival(PFS) | 12 months
Objective response rate(ORR) | baseline, week 6, weeks 12,week 18, week 24
Disease control rate(DCR) | baseline, week 6, weeks 12,week 18, week 24
Phase Ia&Ib: Average change in pain assessed using analgesic medication records per cycle from baseline to each assessment timepoint. | Within 24 weeks from baseline
  Use the analgesic medication record form to document the type, dosage, and frequency of analgesics taken by the subject, thereby evaluating changes in the subject's pain level.

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gagnon B, Murphy J, Simonyan D, Penafuerte CA, Sirois J, Chasen M, Tremblay ML. Cancer anorexia-cachexia syndrome is characterized by more than one inflammatory pathway. J Cachexia Sarcopenia Muscle. 2024 Jun;15(3):1041-1053. doi: 10.1002/jcsm.13430. Epub 2024 Mar 13. PMID 38481033
- [Background] Clamon G, Byrne MM, Talbert EE. Inflammation as a Therapeutic Target in Cancer Cachexia. Cancers (Basel). 2022 Oct 26;14(21):5262. doi: 10.3390/cancers14215262. PMID 36358681
- [Background] Garcia GE, Truong LD, Chen JF, Johnson RJ, Feng L. Adenosine A(2A) receptor activation prevents progressive kidney fibrosis in a model of immune-associated chronic inflammation. Kidney Int. 2011 Aug;80(4):378-88. doi: 10.1038/ki.2011.101. Epub 2011 Apr 20. PMID 21508927
- [Background] Day YJ, Marshall MA, Huang L, McDuffie MJ, Okusa MD, Linden J. Protection from ischemic liver injury by activation of A2A adenosine receptors during reperfusion: inhibition of chemokine induction. Am J Physiol Gastrointest Liver Physiol. 2004 Feb;286(2):G285-93. doi: 10.1152/ajpgi.00348.2003. PMID 14715520
- [Background] Zhang H, Garcia JM. Anamorelin hydrochloride for the treatment of cancer-anorexia-cachexia in NSCLC. Expert Opin Pharmacother. 2015 Jun;16(8):1245-53. doi: 10.1517/14656566.2015.1041500. Epub 2015 May 6. PMID 25945893
- [Background] Mochamat, Cuhls H, Marinova M, Kaasa S, Stieber C, Conrad R, Radbruch L, Mucke M. A systematic review on the role of vitamins, minerals, proteins, and other supplements for the treatment of cachexia in cancer: a European Palliative Care Research Centre cachexia project. J Cachexia Sarcopenia Muscle. 2017 Feb;8(1):25-39. doi: 10.1002/jcsm.12127. Epub 2016 Jul 20. PMID 27897391
- [Background] Anderson LJ, Albrecht ED, Garcia JM. Erratum to: Update on Management of Cancer-Related Cachexia. Curr Oncol Rep. 2017 Mar;19(3):22. doi: 10.1007/s11912-017-0595-4. No abstract available. PMID 28293870
- [Background] Dev R, Wong A, Hui D, Bruera E. The Evolving Approach to Management of Cancer Cachexia. Oncology (Williston Park). 2017 Jan 15;31(1):23-32. PMID 28090619
- [Background] Kimura M, Naito T, Kenmotsu H, Taira T, Wakuda K, Oyakawa T, Hisamatsu Y, Tokito T, Imai H, Akamatsu H, Ono A, Kaira K, Murakami H, Endo M, Mori K, Takahashi T, Yamamoto N. Prognostic impact of cancer cachexia in patients with advanced non-small cell lung cancer. Support Care Cancer. 2015 Jun;23(6):1699-708. doi: 10.1007/s00520-014-2534-3. Epub 2014 Nov 29. PMID 25430482
- [Background] Takayama K, Atagi S, Imamura F, Tanaka H, Minato K, Harada T, Katakami N, Yokoyama T, Yoshimori K, Takiguchi Y, Hataji O, Takeda Y, Aoe K, Kim YH, Yokota S, Tabeta H, Tomii K, Ohashi Y, Eguchi K, Watanabe K. Quality of life and survival survey of cancer cachexia in advanced non-small cell lung cancer patients-Japan nutrition and QOL survey in patients with advanced non-small cell lung cancer study. Support Care Cancer. 2016 Aug;24(8):3473-80. doi: 10.1007/s00520-016-3156-8. Epub 2016 Mar 22. PMID 27003901
- [Background] Jain R, Handorf E, Khare V, Blau M, Chertock Y, Hall MJ. Impact of Baseline Nutrition and Exercise Status on Toxicity and Outcomes in Phase I and II Oncology Clinical Trial Participants. Oncologist. 2020 Feb;25(2):161-169. doi: 10.1634/theoncologist.2019-0289. Epub 2019 Nov 20. PMID 32043776
- [Background] Baracos VE, Martin L, Korc M, Guttridge DC, Fearon KCH. Cancer-associated cachexia. Nat Rev Dis Primers. 2018 Jan 18;4:17105. doi: 10.1038/nrdp.2017.105. PMID 29345251
- [Background] Scherbakov N, Doehner W. Cachexia as a common characteristic in multiple chronic disease. J Cachexia Sarcopenia Muscle. 2018 Dec;9(7):1189-1191. doi: 10.1002/jcsm.12388. Epub 2019 Jan 13. No abstract available. PMID 30637985
- [Background] Fearon K, Strasser F, Anker SD, Bosaeus I, Bruera E, Fainsinger RL, Jatoi A, Loprinzi C, MacDonald N, Mantovani G, Davis M, Muscaritoli M, Ottery F, Radbruch L, Ravasco P, Walsh D, Wilcock A, Kaasa S, Baracos VE. Definition and classification of cancer cachexia: an international consensus. Lancet Oncol. 2011 May;12(5):489-95. doi: 10.1016/S1470-2045(10)70218-7. Epub 2011 Feb 4. PMID 21296615
- [Background] Arends J, Bachmann P, Baracos V, Barthelemy N, Bertz H, Bozzetti F, Fearon K, Hutterer E, Isenring E, Kaasa S, Krznaric Z, Laird B, Larsson M, Laviano A, Muhlebach S, Muscaritoli M, Oldervoll L, Ravasco P, Solheim T, Strasser F, de van der Schueren M, Preiser JC. ESPEN guidelines on nutrition in cancer patients. Clin Nutr. 2017 Feb;36(1):11-48. doi: 10.1016/j.clnu.2016.07.015. Epub 2016 Aug 6. PMID 27637832